CLINICAL TRIAL: NCT00347438
Title: A Phase II Study to Evaluate the Efficacy, Safety, and Genomic Markers of Response of Capecitabine as NeoAdjuvant Therapy in Women With Newly Diagnosed Locally Advanced Breast Cancer
Brief Title: Capecitabine as NeoAdjuvant Therapy in Locally Advanced Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: a result of slow accrual
Sponsor: University of Chicago (Other)
Collaborators: Breast Cancer Research Foundation (Other); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14201B
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer
Keywords: breast cancer; neoadjuvant; locally advanced
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capecitabine (Experimental): Capecitabine will be given at 1000mg/m2 twice daily for 2 weeks x 8 cycles, with a one-week pause in-between cycles.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Capecitabine twice daily for 14 days followed by 7 days without taking drug (1 cycle). This schedule is followed for 8 cycles (about 24 weeks).
  Other Names: Xeloda

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of capecitabine before surgery.

The study will also help gain more information about the effects of the capecitabine on physical and emotional well-being and how well the participants on capecitabine follow the study drug plan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced, histologically confirmed adenocarcinoma of the female breast. Women with ulcerated breast lesions may be enrolled. Patients with asymptomatic metastases to the bone are eligible.
* Ability to provide written informed consent prior to study-specific screening procedures
* TNM Stage:T3-4, N0-3 M0; Patients with asymptomatic bone metastases may be enrolled. Patients with large T2 tumors whose surgeons believe their results with breast conserving surgery will be improved by neoadjuvant therapy may be enrolled.
* Age 18 years or older
* Negative serum or urine pregnancy test within 7 days prior to starting therapy (female patients of childbearing potential).
* Performance status 0-1
* Required Initial Laboratory Data:
* Granulocytes >=1,200/µl
* Platelet count >=100,000/µl
* Calculated Creatinine Clearance > 30 mL/min
* Total bilirubin <= Upper Limit Normal
* Alkaline Phosphatase <=Upper Limit Normal
* SGPT, SGOT <=Upper Limit Normal
* Normal chest x-ray

Exclusion Criteria:

* HER2 positive breast cancer
* Pregnant or lactating woman
* Life expectancy < 3 months
* Serious, uncontrolled, concurrent infection(s)
* Any prior fluoropyrimidine therapy or other chemotherapy
* Prior unanticipated severe reaction to fluoropyrimidine therapy, or known hyper-sensitivity to 5-fluorouracil or known DPD deficiency.
* Patients who have received more than four weeks of tamoxifen therapy for this malignancy.
* Treatment for other carcinomas within the last five years, except cured non- melanoma skin and treated in-situ cervical cancer.
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
* Evidence of metastatic disease to sites other than the bone or with symptomatic bone lesions.
* Other serious uncontrolled medical conditions that the investigator feels might compromise study participation.
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
* Known, existing uncontrolled coagulopathy or concurrent treatment with Coumadin and Phenytoin
* Any of the following laboratory values:
* Abnormal hematologic values (neutrophils < 1.0 x 109/L, platelet count < 100 x 109/L)
* Impaired renal function (estimated creatinine clearance <30ml/min as calculated with Cockcroft-Gault equation)
* Serum bilirubin > upper normal limit.
* SGOT, SGPT > upper normal limit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olufunmilayo I Olopade, MD, Principal Investigator — University of Chicago
Locations (3):
- University of Chicago, Chicago, Illinois, United States
- Nigeria (2):
  - University of Ibadan, Ibadan
  - Obafemi Awolowo University, Ile-Ife

RESULTS

PARTICIPANT FLOW:
Groups:
- Capecitabine: Planned treatment consisted of 24 weeks of capecitabine at a dose of 1000 mg/m^2 twice daily.
Period: Overall Study
Arm/Group | Capecitabine
Started | 18
Completed | 16
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Capecitabine
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Clinical Response Rate (OCR)
Description: Overall clinical response rate (OCR) was defined as a proportion of patients with a best response of Complete Clinical Response (CCR) or Partial Clinical Response (PCR). CCR was defined as complete disappearance of all measurable malignant disease, and no new malignant lesion, disease-related symptoms, or evidence of evaluable disease. PCR was defined as reduction by at least 50% of the sum of the products of the longest perpendicular diameters of all measurable lesions.
Time Frame: After the first three cycles of therapy, an average of 9 weeks
Population: This study was terminated early as a result of slow accrual. Thus, outcome measures were reported only for 16 patients who completed the first three cycles of capecitabine chemotherapy.
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine
Number analyzed (Participants) | 16
percentage of participants | 31.3

2. Primary Outcome: Partial Clinical Response Rate (PR)
Description: Partial Clinical Response (PR) was defined as reduction by at least 50% of the sum of the products of the longest perpendicular diameters of all measurable lesions.
Time Frame: After the first three cycles of therapy, an average of 9 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Capecitabine
Number analyzed (Participants) | 16
participants | 5

3. Primary Outcome: Complete Clinical Response Rate (CCR)
Description: Complete Clinical Response (CCR) was defined as complete disappearance of all measurable malignant disease, and no new malignant lesion, disease-related symptoms, or evidence of evaluable disease.
Time Frame: After the first three cycles of therapy, an average of 9 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine
Number analyzed (Participants) | 16
percentage of participants | 0

4. Primary Outcome: Complete Pathologic Response Rate (cPR)
Description: Complete Pathologic Response rate (cPR) was defined as the absence of invasive breast cancer in the breast (mastectomy or lumpectomy) specimen at the time of definitive surgery.
Time Frame: After the first three cycles of therapy, an average of 9 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine
Number analyzed (Participants) | 16
percentage of participants | 0

ADVERSE EVENTS:
Arm/Group | Capecitabine
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 15/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine (N=16)
Diarrhea (Gastrointestinal disorders) | 3
Skin rash (Skin and subcutaneous tissue disorders) | 1
Hand and foot syndrome (Skin and subcutaneous tissue disorders) | 12
Fatigue (General disorders) | 1
Dizziness (Nervous system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes